CLINICAL TRIAL: NCT02494674
Title: Using Bite Counter for Weight Loss: A One-month Usability Trial to Test the Effectiveness of Using a Wearable Bite Counter to Assist With Dietary Self-monitoring
Brief Title: Using Bite Counter for Weight Loss: A One-month Usability Trial to Test the Effectiveness of Using the Bite Counter
Acronym: Bites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00036795
Record Dates: First submitted 2015-07-06; First posted 2015-07-10 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bite Counter tracking (Experimental): Study participants will be asked to track their energy intake via a wearable device called the Bite Counter. Participants will attend weekly meetings to provide feedback on the Bite Counter.
  Interventions: Behavioral: Bite Counter tracking

INTERVENTIONS:
Behavioral: Bite Counter tracking — Participants will be asked to use the bite counter to track all meals and provide feedback on using the bite counter for dietary self-monitoring.

SUMMARY:
This is a 1-month study that will examine the use of podcasting and a wearable wrist-worn device to track calorie intake and promote weight loss. A podcast is a digital audio file that can be listened to on portable media players, like iPods, and personal computers. This study will run from July 14, 2015 to August 11, 2015. In this study, you will receive weight loss information delivered via twice weekly podcasts. You will also track each meal you eat by wearing a provided watch-like device.

DETAILED DESCRIPTION:
This study will last approximately 1 month (about 4 weeks). Participants will need to attend one 1.5-hour orientation meeting, baseline assessment, and training meeting, and then weekly 1-hour meetings for four weeks (5 meetings total). Participants will listen to 2 podcasts per week and will be encouraged to monitor exercise and body weight and track each meal using the provided wearable, wrist worn device. Each of the podcasts will take about 15 - 20 minutes to listen to and so participants should expect to spend 30 - 40 minutes each week listening to podcasts and up to 3 hours completing other study-related activities each week-including attending the weekly meetings-for a total of about 4 hours per week.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* BMI between 25- 49.9 kg/m2
* live in Columbia, South Carolina area
* be able to attend all assessment visits
* have access to the Internet, a computer, and a smartphone (iPhone, Android, etc.)
* have MD consent for participation if currently on blood pressure medications, have issues with dizziness, or have bone or joint issues
* be free of an eating disorder as screened by the Eating disorder Screen for Primary care. (If a participant has an eating disorder, they will be referred to their family physician)
* no current participation in a weight loss program or taking weight loss medications (although participants may be trying to lose weight on their own)
* able to prepare all their own meals (i.e. not living on-campus)

Exclusion Criteria:

* major health or psychiatric diseases, drug or alcohol dependency, thyroid conditions, or pregnancy
* pregnant (or have been pregnant in the last 6 months), anticipating on becoming pregnant in the next 7 months, or currently breastfeeding o Women who are pregnant should not be pursuing weight loss and should be under the direct care of a physician. Therefore women who are pregnant or who are anticipating they might be pregnant should not participate in this study. If a woman becomes pregnant during the study, she will be advised to consult her care provider and will be dropped from the weight loss study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Body Weight (kg) | 4 weeks
  Assessed with a digital scale accurate to 0.1 kg

SECONDARY OUTCOMES:
Energy intake (kilocalories) | 4 weeks
  Assessed via 2 unannounced 24-hour dietary recalls

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-McGrievy, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States